CLINICAL TRIAL: NCT03016533
Title: Open-label Access to Dolutegravir for HIV-1 Infected Children and Adolescents Completing IMPAACT Studies P1093 and P2019
Brief Title: Dolutegravir Study in HIV-1 Participants Completing IMPAACT Studies P1093 and P2019
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 205858
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Results first posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: HIV Infections
Keywords: Dolutegravir; Continued access study; HIV-1; ABC/DTG/3TC; Pediatric
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dolutegravir (DTG) (Experimental): Participants that received DTG film-coated tablets or film-coated dispersible tablets in the parent study P1093, at appropriate doses selected as per their age and weight bands.
  Interventions: Drug: Dolutegravir film-coated tablets; Drug: Dolutegravir film-coated dispersible tablets
- Abacavir/Dolutegravir/Lamivudine(ABC/DTG/3TC) (Experimental): Participants that received ABC/DTG/3TC immediate release tablets or film-coated dispersible tablets in the parent study P2019, at appropriate doses selected as per their age and weight bands.
  Interventions: Drug: ABC/DTG/3TC immediate release tablets; Drug: ABC/DTG/3TC film-coated dispersible tablets

INTERVENTIONS:
Drug: Dolutegravir film-coated tablets — Dolutegravir film-coated tablets will be provided as 50 mg tablets.
  Arms: Dolutegravir (DTG)
Drug: Dolutegravir film-coated dispersible tablets — Dolutegravir film-coated dispersible tablets will be provided as 5 mg dispersible tablets. It will be administered at the appropriate dose as determined by results of the parent protocol to participants as per their age and weight band.
  Arms: Dolutegravir (DTG)
Drug: ABC/DTG/3TC immediate release tablets — ABC/DTG/3TC immediate release tablets will be provided as biconvex, oval tablets containing 600 mg ABC, 50 mg DTG and 300 mg 3TC.
  Arms: Abacavir/Dolutegravir/Lamivudine(ABC/DTG/3TC)
Drug: ABC/DTG/3TC film-coated dispersible tablets — ABC/DTG/3TC dispersible tablets will be provided as biconvex, oval, film-coated tablets containing 60 mg ABC, 5 mg DTG and 30 mg 3TC.
  Arms: Abacavir/Dolutegravir/Lamivudine(ABC/DTG/3TC)

SUMMARY:
Dolutegravir is a potent integrase strand transfer inhibitor. Abacavir/dolutegravir/lamivudine (ABC/DTG/3TC) is a fixed dose combination regimen containing two nucleoside reverse transcriptase inhibitors and dolutegravir. This is a phase 3b, non-randomized, open-label, multi-center, two treatment rollover study. The primary objective of this pediatric interventional study is to provide continued access to age appropriate formulations of investigational product (dolutegravir), either as Tivicay or as part of fixed dose combination ABC/DTG/3TC, for eligible participants who previously participated in parent studies P1093 (NCT01302847) or P2019 (NCT03760458) and who cannot locally access age appropriate formulations of dolutegravir or ABC/DTG/3TC in the public sector. The P1093 study was designed to evaluate the pharmacokinetics (PK), safety, tolerability and antiviral activity of dolutegravir in combination with optimized background regimens in human immunodeficiency virus type 1 (HIV-1) experienced adolescents and children as well as treatment naïve infants and toddlers. The P2019 study was designed to evaluate PK, safety, tolerability and antiviral activity of ABC/DTG/3TC dispersible and immediate release tablets in HIV-1-infected children. Participants who have tolerated investigational product in the parent studies without any significant toxicity or signs of virologic failure leading to the permanent discontinuation of investigational product and withdrawal from the parent study will be considered for this open label continued access study. Participants will receive their age/weight appropriate dose of investigational product as defined in the parent study. The duration of participation in the study will extend until age appropriate formulations of Tivicay or ABC/DTG/3TC receive local (by country) regulatory approval and are available in those countries from another source (e.g. government programs, aid programs, assistance programs, etc.) or the participant is no longer deriving benefit from treatment or meets a protocol defined reason for discontinuation. Participants will be enrolled after all screening procedures have been completed. In most cases, the Screening visit will overlap with the participants penultimate visit on the parent study (at Week 180 of P1093, or Week 36 of the P2019 study). Participants who meet all entry criteria may enroll and will be seen in the clinic every 12 weeks for a safety evaluation and to receive investigational product. It is estimated that no more than 300 participants will be enrolled in this study. Tivicay is a registered trademark of ViiV Healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have completed participation in one of the following parent studies, for the duration noted, with continued benefit from investigational product:

  1. P1093 parent study through at least Week 180;
  2. P2019 parent study through at least Week 48.
* Participant with evidence of Virological Failure in either parent study must have eligibility for this rollover study discussed and agreed with the ViiV Healthcare Medical Monitor.
* Virological control:

  1. Participants in parent study P1093 must have virological control defined as HIV-1 ribonucleic acid (RNA) <400 copies per milliliter (c/mL) at their penultimate visit (on or after the Week 180 visit);
  2. Participants in parent study P2019 must have virological control defined as HIV-1 RNA <200 c/mL at their penultimate visit (on or after Week 36).
* Evidence of continued benefit from IP during the subject's participation in the parent study (P1093 or P2019)

  1. At screening, Investigators will submit a clinical summary verifying evidence of continued benefit from IP during the subject's participation in the parent study (P1093 or P2019).
  2. The summary will be submitted via the PPD ePIP system to the Study Medical Monitor who will review and confirm if the inclusion criterion has been met.
  3. Confirmation from the Study Medical Monitor is required to meet this eligibility criterion
* Males and Females: All participants who are engaging in sexual activity should be counseled on safer sexual practices including the use and benefit/risk of effective barrier methods (example [e.g.] male condom) and on the risk of HIV transmission to an uninfected partner. Females: Female participants who are of child- bearing potential and who are engaging in sexual activity that could lead to pregnancy, must agree to use one of the acceptable birth control methods until the last dose of study medication and completion of the follow-up visit (4 weeks after the last dose). Condoms are recommended in addition, because their appropriate use is the only contraception method effective for preventing HIV-1 transmission.
* Parent or legal guardian or participant >=18 years of age is able and willing to provide signed informed consent.

Exclusion Criteria:

* Confirmed virologic failure with evidence of resistance to:

  1. DTG in the P1093 parent study, or
  2. ABC, DTG or 3TC (with the exception of M184V) in the P2019 parent study
* Presence of any active AIDS defining opportunistic infection.
* Known >=grade 3 laboratory toxicities prior to study entry (e.g. neutrophil count, hemoglobin, platelets, aspartate aminotransferase [AST], alanine aminotransferase [ALT], lipase, serum creatinine and total bilirubin) would be considered exclusionary if identified at or after the penultimate parent study visit, prior to enrollment in the study... Repeat testing is allowed for eligibility determination.
* Previous permanent discontinuation from investigational product in the parent study due to toxicity, intolerance or pregnancy.
* Known ALT >=5 times the upper limit of normal (ULN), or ALT >=3 times ULN and bilirubin >=1.5 times ULN (with >35 percent [%] direct bilirubin) would be considered exclusionary if identified at or after the penultimate parent study visit, prior to enrolment in the study.. Participants with moderate to severe hepatic impairment (Class B or greater) as determined by Child-Pugh classification should be excluded.
* Participants positive for hepatitis B virus at any time prior to entry (hepatitis B virus surface antigen positive).
* Females who are pregnant or plan to become pregnant or breastfeed during the study.
* Participant is currently participating in or has participated in a study with a compound or device that is not commercially available within 30 days of signing informed consent, unless permission from the sponsor's medical monitor is granted.
* Presence of any history of allergy/sensitivity to any of the study drugs.
* Participants transitioning from the P2019 study (taking ABC/DTG/3TC) have evidence of being Human Leukocyte Antigen-B*5701- positive based on documented testing at any time prior to entry.
* Use of any disallowed medications at time of Screening.
* Anticipated need for Hepatitis C virus therapy with interferon or any drugs that have potential for adverse drug: drug interactions with study treatment throughout the entire study period.
* Participant is unlikely to adhere to the study procedures, keep appointments, or is planning to relocate during the study.
* Clinical or symptomatic evidence of pancreatitis, as determined by the clinician.
* Any condition (including but not limited to alcohol and drug use) that would, in the opinion of the site investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2024-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (17):
- United States (3):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Memphis, Tennessee
- GSK Investigational Site, Gaborone, Botswana
- Brazil (4):
  - GSK Investigational Site, Belo Horizonte
  - GSK Investigational Site, Nova Iguaçu
  - GSK Investigational Site, RibeirAo PretoSP
  - GSK Investigational Site, Rio de Janeiro
- South Africa (4):
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Soweto
  - GSK Investigational Site, Umlazi
- GSK Investigational Site, Moshi, Tanzania
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Chiang Rai
- GSK Investigational Site, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Study sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed one of the parent studies, either P1093 (NCT01302847) or P2019 (NCT03760458), were enrolled in this rollover study. Participants entered and were evaluated in the study at various study sites beginning June 2017 through December 2024.
Period: Overall Study
Arm/Group | Dolutegravir (DTG) | Abacavir/Dolutegravir/Lamivudine(ABC/DTG/3TC)
Started | 61 | 39
Completed | 53 | 29
Not Completed | 8 | 10
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 5 | 10
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dolutegravir (DTG) | Abacavir/Dolutegravir/Lamivudine(ABC/DTG/3TC) | Total
Number analyzed (Participants) | 61 | 39 | 100
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 7.5 (4.07) | 6.7 (3.14) | 7.2 (3.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 17 | 49
  Male | 29 | 22 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN | 11 | 15 | 26
  BLACK OR AFRICAN AMERICAN | 47 | 23 | 70
  WHITE | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Continued Access to Age Appropriate Formulation of Dolutegravir
Time Frame: From Day 1 (rollover visit from the parent study) through Year 7 (end of study) or early withdrawal
Population: The analysis was performed on the Safety Set, which included all participants who received at least one dose of study intervention once enrolled in the study. The presented number is representing participants that completed all visits in parent studies.
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir (DTG) | Abacavir/Dolutegravir/Lamivudine(ABC/DTG/3TC)
Number analyzed (Participants) | 61 | 39
Participants | 53 | 29

2. Secondary Outcome: Number of Participants With Any Serious Adverse Events (SAEs)
Description: An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, results in abnormal pregnancy outcomes or any other situation based on appropriate medical or scientific judgement. Any = occurrence of the event regardless of intensity grade or relationship to the study interventions.
Time Frame: From Day 1 (rollover visit from the parent study) through Year 7 (end of study) or early withdrawal
Population: The analysis was performed on the Safety Set, which included all participants who received at least one dose of study intervention once enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir (DTG) | Abacavir/Dolutegravir/Lamivudine(ABC/DTG/3TC)
Number analyzed (Participants) | 61 | 39
Participants | 5 | 3

3. Secondary Outcome: Number of Participants With SAEs Leading to Discontinuation of Study Treatment
Time Frame: From Day 1 (rollover visit from the parent study) through Year 7 (end of study) or early withdrawal
Population: The analysis was performed on the Safety Set .
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir (DTG) | Abacavir/Dolutegravir/Lamivudine(ABC/DTG/3TC)
Number analyzed (Participants) | 61 | 39
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Any Clinical or Laboratory Adverse Events (AEs) Leading to Discontinuation of Study Treatment
Time Frame: From Day 1 (rollover visit from the parent study) through Year 7 (end of study) or early withdrawal
Population: The analysis was performed on the Safety Set .
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir (DTG) | Abacavir/Dolutegravir/Lamivudine(ABC/DTG/3TC)
Number analyzed (Participants) | 61 | 39
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs and AEs leading to study intervention discontinuation were collected from Day 1 (rollover visit from the parent study) through Year 7 (end of study) or early withdrawal.
Arm/Group | Dolutegravir (DTG) | Abacavir/Dolutegravir/Lamivudine(ABC/DTG/3TC)
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/39
Serious Adverse Events (participants affected / at risk) | 5/61 | 3/39
Other Adverse Events (participants affected / at risk) | 0/61 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dolutegravir (DTG) (N=61) | Abacavir/Dolutegravir/Lamivudine(ABC/DTG/3TC) (N=39)
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT03016533/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT03016533/SAP_001.pdf